CLINICAL TRIAL: NCT00598871
Title: A Randomized, Double-Mask, Placebo-Controlled, Dose Response, Phase 2 Study of the Safety and Efficacy of Thymosin Beta 4 in the Treatment of Diabetic Patients' Corneal Wounds Resulting From Epithelial Debridement During Vitrectomy
Brief Title: A Phase 2 Study of the Safety and Efficacy of Thymosin Beta 4 for Treating Corneal Wounds
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: ReGenTree, LLC (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGN-DV-201
Record Dates: First submitted 2007-12-19; First posted 2008-01-23 (Estimated); Results first posted 2010-04-13 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes
Keywords: Thymosin beta 4; Corneal wound healing; Vitrectomy; Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — thymosin beta(4)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): There are 2 groups: active drug and placebo. The patients in the placebo arm receive an administration of eyedrops to the affected eye, identical to the active drug but with no thymosin beta 4 (0.00% thymosin beta 4, w/w), 2 drops 4 times a day (breakfast, lunch, dinner, and bedtime) for 14 days. The first of 4 daily doses will be administered following surgery (vitrectomy).
  Interventions: Other: Placebo
- 1 (Active Comparator): There are 2 groups: active drug and placebo. The patients in the active comparator arm receive an administration of 0.01% Tβ4 (w/w) eyedrops to the affected eye, 2 drops 4 times a day (breakfast, lunch, dinner, and bedtime) for 14 days. The first of 4 daily doses will be administered following surgery (vitrectomy).
  Interventions: Drug: Thymosin Beta 4 (Tβ4)

INTERVENTIONS:
Drug: Thymosin Beta 4 (Tβ4) — There are 2 groups: active drug and placebo. The patients in the active arm receive an administration of 0.01% Tβ4 (w/w) eyedrops to the affected eye, 2 drops 4 times daily (breakfast, lunch, dinner, and bedtime) for 14 days. The first of 4 daily doses will be administered following surgery (vitrectomy).
  Other Names: Thymosin Beta 4 eye drops; Tβ4 eye drops; RGN-259
  Arms: 1
Other: Placebo — There are 2 groups: active drug and placebo. The patients in the placebo arm receive an administration of 0.00% Tβ4(w/w) eyedrops to the affected eye, 2 drops four times a day (QID) (breakfast, lunch, dinner, and bedtime) for 14 days. The first of 4 daily doses will be administered following surgery (vitrectomy).
  Arms: 2

SUMMARY:
As a consequence of damage to multiple organ systems throughout the course of their disease, diabetic patients suffer a number of chronic complications giving rise to increased morbidity, mortality, and health care costs specific to this population. Within the ophthalmic domain, diabetic retinopathy (DR) frequently induces serious visual impairment. Although DR can be addressed surgically, surgery remains a less than ideal intervention within this population with a well-characterized compromised ability to heal. The introduction of a therapeutic agent that could accelerate wound closure and decrease healing time, thereby reducing the risk and incidence of infection and corneal scarring in these susceptible patients, would represent a significant clinical and pharmacoeconomic advance in the treatment of this condition.

DETAILED DESCRIPTION:
In individuals with certain clinical conditions, such as diabetes, corneal epithelial defects persist and do not necessarily respond to conventional treatment regimens because of delayed epithelial wound healing. While wound closure should occur following an injury to the corneal epithelium, a timely re-establishment of the epithelial barrier is of utmost importance.

The wound repair process is intricately linked to a complex inflammatory response that must be properly regulated to ensure healing and optimal visual outcome. Infiltration of inflammatory cells into injured corneal tissue is a hallmark of wound repair, and the association of polymorphonuclear (PMN) leukocyte infiltration with sterile corneal ulceration is well recognized. Retardation of epithelial recovery by persistent inflammation, release of enzymatic products from degranulating PMN, and stimulation of mononuclear leukocytes by cytokines all contribute to poor re-epithelialization.

It has been shown that diabetic corneas manifest reduced rates of epithelial healing after denudement. Yet, in the diabetic patient, not only is the rate of corneal epithelial healing of clinical concern, abnormalities inherent in the diabetic corneal epithelial cytoarchitecture can cause substantial impediments to normal stromal healing. Histologically, diabetic corneas typically demonstrate thickening of the epithelial basal membrane (BM), decreased number of hemidesmosomes, and decreased number of nerve fiber endings. Studies of BM changes in diabetic corneas have yielded information regarding poor adhesion of the epithelial BM to the stroma. During vitrectomy in diabetic patients, when the cornea epithelium is removed, it separates as an intact sheet and the entire thickened BM, characteristic of diabetes, adheres to the epithelium. In contrast, when normal epithelium is removed by scraping, the BM remains adherent to the stroma.

Because patients with diabetic retinopathy (DR) corneas have delayed wound healing, the expression of thymosin beta 4 (Tβ4) as a potent epithelial cell migration stimulator in DR corneas was investigated. Human DR corneas were analyzed and were found to express significantly less Tβ4 compared to normal corneas, suggesting that the use of Tβ4 may accelerate the wound-healing process in this model.

ELIGIBILITY:
Inclusion Criteria

* Type 1 or Type 2 diabetes mellitus.
* Patients who have an expected minimum 50% likelihood of requiring corneal epithelial debridement in the opinion of the Investigator Size of wound should be 8 mm.
* Signed written informed consent by patient or legal guardian.

Exclusion Criteria

* Have current or history of herpetic eye disease in the past 3 years.
* Display evidence of keratitis.
* Have Sjögren's syndrome.
* Have corneal scarring, opacity, or dystrophy.
* Have a history of malignancy.
* Have a history of HIV or AIDs
* Are pregnant or lactating females.
* Are females who can become pregnant.
* Have a known hypersensitivity to the study drug.
* May be regarded as unreliable for the study.
* Have previously participated in this study.
* Experience any complication during the vitrectomy procedure itself, which will exclude the patient from participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Crockford, Study Director — RegeneRx Biopharmaceuticals, Inc.
Locations (5):
- United States (5):
  - United Medical Research Institute, Inglewood, California
  - Doheny Eye Institute, Los Angeles, California
  - Magruder Eye Institue, Orlando, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Western Carolina Retinal Associates, PA, Asheville, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in January 2008 and ended February 2009 using 4 sites (Hospital Medical Centers). Only the first dose group was completed before suspending the trial due to low patient availability.The procedure of debridement was discontinued in most centers, thus making the availability of surgical subject extremely small.
Pre-assignment Details: Prior to randomization, patients needed to meet specific inclusion and exclusion criteria.There was no run-in period.
Groups:
- Placebo: Administration of 0.00% Thymosin beta 4 (Tβ4) weight/weight(w/w) eyedrops to the affected eye, 2 drops 4 times a day (breakfast, lunch, dinner, and bedtime) for 14 days. The first of 4 daily doses will be administered following surgery (vitrectomy).
- Active Drug: Administration of 0.01% Tβ4 weight/weight (w/w) eyedrops to the affected eye, 2 drops 4 times a day (breakfast, lunch, dinner, and bedtime) for 14 days. The first of 4 daily doses will be administered following surgery (vitrectomy).
Period: Overall Study
Arm/Group | Placebo | Active Drug
Started | 3 | 9
Completed | 3 | 8
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Active Drug | Total
Number analyzed (Participants) | 3 | 9 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (3.1) | 51.4 (15.0) | 49.4 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) After Treatment With Thymosin Beta 4 in the Target Eye of Diabetic Patients During Vitrectomy
Description: Number of participants with Number of Treatment Emergent Adverse Events (TEAEs) in the Target Eye in diabetic patients who had undergone epithelial debridement during vitrectomy and treated with thymosin beta 4
Time Frame: 14 days
Population: Intent to Treat (ITT), Last Observation Carried Forward (LOCF)
Measure: Number; unit: Participants
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 3 | 9
Participants | 3 | 9

2. Secondary Outcome: Number of Participants With Corneal Epithelial Wound Healing at Day 14 (End of Treatment)
Description: Number of diabetic patients who had undergone epithelial debridement during vitrectomy resulted in complete corneal wound closure of the affected eye at the end of treatment (Day 14)
Time Frame: 14 days
Population: Analysis per protocol, ITT (Intent to treat), using LOCF (Last Observation Carried Over)
Measure: Number; unit: participants
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 3 | 9
participants | 3 [29.2 to 100] | 9 [66.4 to 100]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected on a daily basis for the first 14 days and during follow-up at Day 28
Description: AEs were collected daily
Arm/Group | Placebo | Active Drug
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/9
Other Adverse Events (participants affected / at risk) | 3/3 | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=3) | Active Drug (N=9)
Anterior Chamber Cells (Eye disorders) | 3 (3) | 6 (6)
Anterior Chamber Flare (Eye disorders) | 3 (3) | 6 (6)
Conjunctival Haemorrhage (Eye disorders) | 2 (2) | 7 (7)
Conjunctival oedema (Eye disorders) | 1 (1) | 6 (6)
Punctate Keratitis (Eye disorders) | 2 (2) | 5 (5)
Corneal disorder (Eye disorders) | 2 (2) | 4 (4)
Corneal oedema (Eye disorders) | 2 (2) | 4 (4)
Eye Pain (Eye disorders) | 0 (0) | 4 (4)
Corneal Erosion (Eye disorders) | 1 (1) | 2 (2)
Eyelid oedema (Eye disorders) | 0 (0) | 3 (3)
Anterior Chamber Fibrin (Eye disorders) | 1 (1) | 1 (1)
Corneal Staining (Investigations) | 2 (2) | 4 (4)
Intraocular Pressure Increased (Investigations) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Anterior Chamber Inflammation (Eye disorders) | 0 (0) | 1 (1)
Corneal epithelium defect (Eye disorders) | 0 (0) | 1 (1)
Corneal Opacity (Eye disorders) | 0 (0) | 1 (1)
Corneal striae (Eye disorders) | 0 (0) | 1 (1)
Eye oedema (Eye disorders) | 0 (0) | 1 (1)
Iris adhesions (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Ocular Discomfort (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Spatial pain (General disorders) | 0 (0) | 1 (1)
Post procedural oedema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
RegeneRx (the Sponsor) agreements may vary with individual investigators, but will not prohibit any investigator from publishing. RegeneRx supports the publication of results from all centers of a multi-center trial but requests that reports based on a single-site data not precede the primary publication of the entire clinical trial.